CLINICAL TRIAL: NCT02493114
Title: Physical Functioning Throughout Lung Cancer Treatment
Acronym: LUCAT
Status: Completed | Type: Observational
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Chris Burtin, Dr, Hasselt University
Other Study IDs: 1
Record Dates: First submitted 2015-06-11; First posted 2015-07-09 (Estimated); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer; Exercise Capacity; Physical Activity; Quality of Life
MeSH Terms: conditions — Lung Neoplasms; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Patients with lung cancer: No study intervention
- Healthy controls: No study intervention

SUMMARY:
This trial investigates the impact of lung cancer treatment on physical status, symptoms and quality of life. Furthermore this trial investigates possible underlying causes and consequences of deconditioning.

DETAILED DESCRIPTION:
Preliminary evidence suggests that patients with lung cancer experience a decrease of exercise tolerance and muscle strength during the course of their treatment. The underlying mechanisms and impact of this change has not yet been investigated. In light of this, our trial will prospectively follow a convenience sample of 150 patients with lung cancer who are undergoing treatment. Patients will be assessed before, during and at the end of the treatment (surgery and/or chemotherapy and/or radiotherapy and/or immunotherapy). The aims of the study are to

1. Investigate physical status, before start of treatment in lung cancer patients in comparison with healthy controls (primary outcome).
2. Investigate changes in physical status over the course of treatment in lung cancer patients (primary outcome).
3. Investigate the relationship between changes in physical status with physical activity and symptoms during treatment for lung cancer (secondary outcome).
4. Investigate the relationship between physical status after treatment for lung cancer and comorbidities, hospitalizations and cancer-related and all-cause mortality (exploratory outcome).

ELIGIBILITY:
Inclusion Criteria:

* undergoing treatment (surgery, chemotherapy, immunotherapy, radiotherapy, and combination of the previous ones)
* WHO performance status of maximal 2

Exclusion Criteria:

* presence of other neoplasms in the last 2 years
* bone metastasis
* progressive neuromuscular and neurological diseases
* unstable cardiac disease
* pulmonary hypertension
* interstitial lung disease
* orthopedic conditions that significantly impair functional status
* mental or psychiatric disorders that impair the ability to comply with study procedures.
* a history of cerebrovascular accident with remaining functional consequences
* a history of lung cancer
* difficulties in understanding and speaking Dutch

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients with a primary diagnosis of non-small-cell lung cancer who will undergo treatment (surgery, chemotherapy, immunotherapy, radiotherapy, and combination of the previous ones) and score a maximal of 2 on the WHO performance status classification, will be eligible for inclusion.
  Healthy matched volunteers will carry out the same assessments once.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2015-07; Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
6MWT | Before start of treatment versus 3 months after treatment initiation
1-minute sit to stand test | Before start of treatment versus 3 months after treatment initiation
SPPB | Before start of treatment versus 3 months after treatment initiation

SECONDARY OUTCOMES:
Handgrip strength | Before start of treatment vs. 3 months after treatment initiation
Daily physical activity (self-reported and accelerometer) | Before start of treatment vs. during treatment (surgery: during hospitalization; radio: week 2; chemo: beginning of cycle 2 and cycle 4 (each cycle is 3 weeks); immuno: beginning of cycle 2 and cycle 4) vs. 3 months after treatment initiation
Quadriceps strength (isometric and isokinetic) | Before start of treatment vs. 3 months after treatment initiation
Respiratory muscle strength (maximal inspiratory and expiratory pressure) | Before start of treatment vs. 3 months after treatment initiation

OTHER OUTCOMES:
Comorbidities | Before start of treatment
Number of hospital admissions | 12 months after treatment initiation
All cause and cancer-related mortality | 12 months after treatment initiation
Symptoms (Visual analogue scales) | Before start of treatment vs. during treatment (surgery: during hospitalization; radio: week 2; chemo: beginning of cycle 2 and cycle 4 (each cycle is 3 weeks); immuno: beginning of cycle 2 and cycle 4) vs. 3 months and 1 year after treatment initiation
Cancer-specific Quality of life (European Organization for the Research and Treatment of Cancer Questionnaire and lung cancer module - EORTC QLQ-C30-LC13) | Before start of treatment vs. during treatment (surgery: during hospitalization; radio: week 2; chemo: beginning of cycle 2 and cycle 4 (each cycle is 3 weeks); immuno: beginning of cycle 2 and cycle 4) vs. 3 months an after treatment initiation
General Health Status (12-item Short Form Health Survey - SF-12) | Before start of treatment vs. 3 months after treatment initiation
General Health Status (EuroQol 5-dimensions) | Before start of treatment vs. during treatment (surgery: during hospitalization; radio: week 2; chemo: beginning of cycle 2 and cycle 4 (each cycle is 3 weeks); immuno: beginning of cycle 2 and cycle 4) vs. 3 and 1 year months after treatment initiation
Daily functioning (Instrumental Activities of Daily Living Scale - IADLS) | Before start of treatment vs. during treatment (surgery: during hospitalization; radio: week 2; chemo: beginning of cycle 2 and cycle 4 (each cycle is 3 weeks); immuno: beginning of cycle 2 and cycle 4) vs. 3 months after treatment initiation
Fatigue (Multidimensional Fatigue Inventory - MFI-20) | Before start of treatment vs. during treatment (surgery: during hospitalization; radio: week 2; chemo: beginning of cycle 2 and cycle 4 (each cycle is 3 weeks); immuno: beginning of cycle 2 and cycle 4) vs. 3 months and 1 year after treatment initiation
Dyspnea (modified medical research council scale - MMRC) | Before start of treatment vs.3 months after treatment initiation
Anxiety and depression (Hospital Anxiety and Depression Scale) | Before start of treatment vs. 3 months after treatment initiation
Care needs (Care Dependency Scale) | Before start of treatment vs. 3 months after treatment initiation
Dyspnea (San Diego Shortness of Breath Questionnaire (SOBQ)) | Before start of treatment vs. during treatment (surgery: during hospitalization; radio: week 2; chemo: beginning of cycle 2 and cycle 4 (each cycle is 3 weeks); immuno: beginning of cycle 2 and cycle 4) vs. 3 months and 1 year after treatment initiation
Depressive symptomatology (Center for Epidemiologic Studies Depression scale (CES-D)) | Before start of treatment vs. 3 months after treatment initiation

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium

REFERENCES:
- [Derived] Quadflieg K, Arents E, Haesevoets S, Van Hulle F, Hermans F, Criel M, Daenen M, Derom E, Spruit MA, Surmont V, Stevens D, Ruttens D, Demeyer H, Burtin C. Impact of cancer treatment on physical functioning, symptoms and health-related quality of life in patients with non-small cell lung cancer: A longitudinal observational study. Respir Med. 2025 Oct;247:108283. doi: 10.1016/j.rmed.2025.108283. Epub 2025 Jul 31. PMID 40752628